CLINICAL TRIAL: NCT07290803
Title: Atopic Dermatitis Disease Registry of Adult and Adolescent Patients Initiating or Switching Systemic Treatments
Brief Title: This Study is a Non-interventional Disease Registry of Adolescent and Adult Patients With Atopic Dermatitis Who Initiate or Switch Any Systemic Treatment
Acronym: ARMADA-AD
Status: Recruiting | Type: Observational
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Other Study IDs: OBS18388; U1111-1311-1824 (Registry Identifier: ICTRP)
Record Dates: First submitted 2025-11-28; First posted 2025-12-18 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Atopic Dermatitis: This study plans to collect information on adolescent and adult patients with atopic dermatitis who initiate or switch any systemic treatment (eg, biologics, oral Janus kinase [JAK] inhibitors, cyclosporine, azathioprine, methotrexate, mycophenolate mofetil) for AD according to the country-specific prescribing information. During the study, investigators will prescribe medical products for treatment of AD per standard of care (SoC) and per medical judgment.

SUMMARY:
The objectives of this prospective non-interventional study are to characterize the existing unmet needs across the spectrum of atopic dermatitis (AD), enhance the understanding of the patient journey, and evaluate the safety and clinical outcomes of systemic AD treatments in a real-world setting. Additionally, patient-specific factors (such as age, skin color, AD flare triggers, previous treatment responses, comorbid conditions, and the extent and site of lesions) will be assessed to better characterize the impact on the treatment journey across a broad age range and diverse geographic regions.

The study will be conducted across 10 countries in 4 different geographical regions, with a follow-up period of 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged more than or equal to (≥) 12 years at the time of consent.
* Confirmed diagnosis of AD, of any severity, according to the Investigator's assessment as aligned with International Classification of Diseases 10th revision (ICD-10) code of L20.
* Prescribed and scheduled to initiate any systemic treatment for AD (including but not limited to biologics, oral Janus kinase (JAK) inhibitors, cyclosporine, azathioprine, methotrexate, mycophenolate mofetil)
* Signed informed consent for registry participation by the patient or parent/legal representative and assent by the patient appropriate to the patient's age, including willingness to participate in long-term follow-up.

Exclusion Criteria:

* Concurrent participation in an interventional clinical trial that administers an investigational drug that modifies patient care.
* Insufficient understanding of the study by the patient and/or parent/guardian.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with any atopic dermatitis severity will be invited to enroll in the registry after the decision has been made to initiate a new systemic medication for the first time or switch systemic therapies. Inclusion in the registry will not influence a patient's treatment course.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-11-17 (Actual); Primary Completion 2034-01-30 (Estimated); Study Completion 2034-01-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Utilizing Atopic Dermatitis (AD) Treatment | Baseline to up to 60 months
  The number (and percentage) of participants taking AD treatments and treatments per patient will be described.
Duration of Treatment | Baseline to up to 60 months
  The duration of AD treatments will be summarized descriptively.
AD Treatment Sequences | Baseline to up to 60 months
  The ordering of AD treatments will be summarized descriptively.
Number of Participants Initiating AD Treatments with Reasons | Baseline to up to 60 months
  The number (and percentage) of patients initiating AD treatment and reasons for initiation will be summarized descriptively.
Number of Participants Interrupting AD Treatment | Baseline to up to 60 months
  The number (and percentage) of patients interrupting AD treatment and reasons for treatment interruption will be summarized descriptively.
Number of Participants Discontinuing AD Treatment | Baseline to up to 60 months
  The number (and percentage) of patients discontinuing AD treatment and reasons for treatment discontinuation will be summarized descriptively.
Number of Participants Switching AD Treatments | Baseline to up to 60 months
  The number (and percentage) of patients switching AD treatment and reasons for treatment switch will be summarized descriptively.
Number of Participants Augmenting AD treatment | Baseline to up to 60 months
  The number (and percentage) of patients augmenting AD treatment will be summarized descriptively.
Number of Participants Modifying AD Treatment Dose | Baseline to up to 60 months
  The number (and percentage) of patients modifying AD treatment dose, reasons for dose modification, and dosing will be summarized descriptively.
Change from Baseline in Extent and Severity of AD Measured with Eczema Area and Severity Index (EASI) | Baseline to up to 60 months
  Clinical outcomes measured using EASI will be summarized at the start of a treatment episode and each follow-up time point.
Change from Baseline in Extent and Severity of AD Measured with Body Surface Area (BSA) | Baseline to up to 60 months
  Clinical outcomes measured using BSA will be summarized at the start of a treatment episode and each follow-up time point.
Change from Baseline in Extent and Severity of AD Measured with Validated Investigator's Global Assessment for Atopic Dermatitis (vIGA-AD) | Baseline to up to 60 months
  Clinical outcomes measured using vIGA-AD will be summarized at the start of a treatment episode and each follow-up time point.
Change from Baseline in Extent and Severity of AD Measured with Revised Investigator's Global Assessment for Atopic Dermatitis (rIGA-AD) | Baseline to up to 60 months
  Clinical outcomes measured using rIGA-AD will be summarized at the start of a treatment episode and each follow-up time point.
Change in Atopic Dermatitis Control Test (ADCT) from Baseline | Baseline to up to 60 months
  The ADCT is a 6-item patient-reported outcomes instrument with a 7-day recall period to measure AD disease control. Total score ranges from 0 to 24.
Change in Patient Global Impression of Severity (PGIS) from Baseline | Baseline to up to 60 months
  The PGIS is a single item tool used to assess current severity of eczema symptoms, scored on a 5-point scale from 1 = no symptoms to 5 = very severe symptoms.
Change in Itch severity as Measured with the Peak Pruritus Numeric Rating Scale (PP-NRS) from Baseline | Baseline to up to 60 months
  The PP-NRS is a single item 0-10 numeric rating scale assessing peak pruritus (itch) associated with AD during the past 24 hours, with 0 = no itch and 10 = worst itch imaginable.
Change in Skin Pain as Measured with Skin Pain Numeric Rating Scale (SP-NRS) from Baseline | Baseline to up to 60 months
  The SP-NRS is a single item 0-10 numeric rating scale assessing skin pain associated with AD during the past 24 hours, with 0 = no pain and 10 = worst possible pain imaginable.
Change in Sleep Disturbance as Measured with Sleep Disturbance Numeric Rating Scale (SD-NRS) from Baseline | Baseline to up to 60 months
  The SD-NRS is a single item 0-10 numeric rating scale assessing sleep disturbance associated with AD, with 0 being 'no sleep loss related to the symptoms of atopic dermatitis' and 10 being 'I did not sleep at all' due to the symptoms of atopic dermatitis.
Remission of AD | Baseline to up to 60 months
  Total remission of all signs and symptoms of AD will be assessed.

SECONDARY OUTCOMES:
Sociodemographic characteristics of Participants | Baseline
  Demographics characteristics including age, sex, body weight, height, geographic region, education level, employment status, smoking and alcohol status will be collected.
Ethnic Origin in Combination with Fitzpatrick Scale | Baseline
  The Fitzpatrick Skin Type Scale was developed based on an individual's reaction to sun exposure and will be completed by the Investigator. Skin types range from I - VI, with scores of I indicating the palest skin tone with no inherent melanin pigmentation, and VI indicating the darkest skin tone with significant amount of melanin.
Disease characteristics of Participants | Baseline
  History of AD (including date of diagnosis, age of onset, specialty of provider who diagnosed condition), AD morphology, including but not limited to, patches, plaques, prurigo nodules, lichenoid papules, perifollicular papules, nummular lesions, and psoriasiform lesions and family history of AD and comorbidities will be collected.
Change from Baseline in Dermatology-specific Quality of Life Measure with Dermatology Life Quality Index (DLQI) | Baseline to up to 60 months
  DLQI is calculated by summing the score of each question resulting in a maximum score of 30 and a minimum score of 0 (higher scores indicate quality of life is more impaired).
Change from Baseline in Dermatology-specific Quality of Life Measure with Children's Dermatology Life Quality Index (CDLQI) | Baseline to up to 60 months
  The CDLQI is calculated by summing the score of each question resulting in a maximum score of 30 and a minimum score of 0 (higher scores indicate quality of life is more impaired).
Change from Baseline in Burden of Assessment Using Patient Health Questionnaire-9 (PHQ-9) | Baseline to up to 60 months
  PHQ-9 is a 9-item, validated, patient-reported questionnaire to assess depression which scores each of the 9 Diagnostic and Statistical Manual of Mental Disorders-IV criteria as "0" (not at all) to "3" (nearly every day). Possible scores range from 0 to 27 and are classified as 1-4: "minimal depression"; 5-9: "mild depression"; 10-14: "moderate depression"; 15-19: "moderately severe depression"; and 20-27: "severe depression".
Change from Baseline in AD Specific Work and Classroom Productivity and Impairment Assessed Using WPAI+CIQ | Baseline to up to 60 months
  Work Productivity and Activity Impairment plus Classroom Impairment Questions (WPAI+CIQ) is a 10-item, patient-reported, validated questionnaire adapted for AD to measure impairments in work, classroom, and regular daily activities over a 7-day period.
Change from Baseline in Treatment Satisfaction Assessed Using Treatment Satisfaction Questionnaire for Medication (TSQM-9) | Baseline to up to 60 months
  The 14-item TSQM-9 is a generic measure of treatment satisfaction, assessing side effects, effectiveness, convenience and global satisfaction, over the last 2 to 3 weeks, or since the patient has last used it. A lower score indicates lower satisfaction with treatment.
Visits with Specialty of Attending Healthcare Provider and Reason for Visit | Baseline to up to 60 months
  Health care resource utilization including visits with specialty of attending health care provider and reason for visit (example, disease flare-up, regular visit, prescription change, adverse event [AE]) will be assessed.
Hospitalizations for AD | Baseline to up to 60 months
  Hospitalization for AD will be assessed.
Prevalence of Comorbid Atopic Conditions | Baseline to up to 60 months
  Prevalence of comorbid atopic conditions (including but not limited to, asthma, allergic conjunctivitis, allergic rhinitis, eosinophilic esophagitis, nasal polyposis, food allergy, prurigo nodularis, chronic spontaneous urticaria, and rhinoconjunctivitis) and non-atopic conditions (including but not limited to, insomnia, anxiety, attention deficit disorder, depression, major adverse cardiovascular event, cardiovascular disease, skin infection, pulmonary disease, osteoporosis, fractures, contact allergy, and inflammatory conditions) will be assessed.
Incidence of Comorbid Atopic Conditions | Baseline to up to 60 months
  Incidence of comorbid atopic conditions (including but not limited to, asthma, allergic conjunctivitis, allergic rhinitis, eosinophilic esophagitis, nasal polyposis, food allergy, prurigo nodularis, chronic spontaneous urticaria, and rhinoconjunctivitis) and non-atopic conditions (including but not limited to, insomnia, anxiety, attention deficit disorder, depression, major adverse cardiovascular event, cardiovascular disease, skin infection, pulmonary disease, osteoporosis, fractures, contact allergy, and inflammatory conditions) will be assessed.
Change from Baseline in Asthma Control Assessed with Asthma Control Questionnaire-5 (ACQ-5) | Baseline to up to 60 months
  ACQ-5 is a 5-item questionnaire used to assess asthma control [33]. Each question is rated on a 7-point scale (0=no impairment; 6=maximum impairment). The ACQ-5 score is calculated using the mean of the 5 items and ranges between 0 (well controlled asthma) to 6 (extremely poorly controlled asthma). The ACQ-5 will only be completed by patients with comorbid asthma.
Occurrence of Concomitant Medication use for AD and Selected Comorbidities | Baseline to up to 60 months
  The occurrence of concomitant medication use for AD and selected comorbidities at baseline and changes (including reason for change) will be summarized.
Number of Adverse Events (SAEs) | Baseline to up to 60 months
  Number of patients experiencing AEs.
Number of Serious Adverse Events (SAEs) | Baseline to up to 60 months
  Number of patients experiencing SAEs.

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - The Center for Dermatology Clinical Research- Site Number : 8400014, Fremont, California
  - St. Jude Clinical Research- Site Number : 8400049, Doral, Florida
  - Skin Care Physicians of Georgia - Macon- Site Number : 8400034, Macon, Georgia
  - Las Vegas Dermatology- Site Number : 8400002, Las Vegas, Nevada
  - Optima Research Portsmouth- Site Number : 8400032, Portsmouth, New Hampshire
  - Innovate Research - Fort Worth- Site Number : 8400016, Fort Worth, Texas

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org